CLINICAL TRIAL: NCT02345109
Title: Verify the Functions and Efficiency of Transtek (Trade Mark) Body Fat Analyzer, 8 Models
Brief Title: Clinical Trial of Transtek Body Fat Analyzer (GBF-835-N2 & Other 7 Models)
Acronym: 15001Analy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leo Wang (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor-Investigator, Leo Wang, Team Leader, BTS International
Organization: BTS International (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: 15001_Analyzer; BTS15001 (Other: BTSInternational)
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Weight; Body Fat Disorder
Keywords: weight; total body water; body fat; muscle mass; bone mass; BMI; visceral fat; calories
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transtek DUT (Experimental): Which measured by DUT: GBF-835-N2, GBF-835-N2 Plus, LS202-B1, Ls202-B1 Plus, LS206-E1, LS206-E1 Plus, GBF-1251-B1, and GBF-1251-B1 Plus.
  Interventions: Device: Transtek DUT; Device: Reference
- Reference (Experimental): Measured by Reference: TRANSTEK® Glass Body Fat Analyzer GBF-1251-B, Tanita® Body Composition Monitor BC-533.
  Interventions: Device: Transtek DUT; Device: Reference

INTERVENTIONS:
Device: Transtek DUT — Measuring weight, total body water, body fat, muscle mass, bone mass, BMI, visceral fat, and calorie.
  Measure each participants by Transtek DUT.
Device: Reference — Measuring weight, total body water, body fat, muscle mass, bone mass, BMI, visceral fat, and calorie. Measure each participants by Reference.

SUMMARY:
The clinical protocol of the clinical testing of this device:

1. Objective of the test: To verify the functions and efficiency of devices.
2. Test methods and procedures: Comparison Test.
3. Device Under Test (DUT): Transtek Body Fat Analyzer, Model: GBF-835-N2, GBF-835-N2 Plus, LS202-B1, LS202-B1 Plus, LS206-E1, LS206-E1 Plus, GBF-1251-B1, and GBF-1251-B1 Plus.
4. Comparison device: TRANSTEK GBF-1251-B and Tanita BC-533.
5. Study endpoints: DUT and the comparison device are substantial equivalence.
6. Statistical methodology used: Description of statistical methods.

DETAILED DESCRIPTION:
1. Test Purpose:

   The aim of clinical test is to collect BMI, body fat, total body water, muscle mass, bone mass, calorie, and visceral fat reading value which measured by DUT and reference device.
2. Target Subject:

   The subject database shall contain at least 30 male and 30 female subjects and all above 10 years old.
3. Test procedures:

   1. Record the name, age, gender, and height of each subject.
   2. Let subject seated calmly for two minutes before test, dry the feet.
   3. Use device to measure weight, body fat, total body water, bone mass, and muscle mass; record reading value.
   4. For each subject, repeat 3) to get 3 pairs measurements.
   5. Repeat step 1) to 4) for every device (DUT: GBF-835-N2, GBF-835-N2 Plus, LS202-B1, LS202-B1 Plus, LS206-E1, LS206-E1 Plus, GBF-1251-B1, and GBF-1251-B1 Plus; and reference device: GBF-1251-B and BC-533).
   6. Repeat step 1) to 5) for each subject.
4. Note:

   1. No motion and speaking are allowed during the measurement.
   2. All DUT use the same algorithms and contact the patient at the same body locations (feet), and operate on the same frequency.
   3. Test environment: Temperature: 22±1℃; Relative humidity: 40~70%.

ELIGIBILITY:
Inclusion Criteria:

* Male, female

Exclusion Criteria:

* Below 10 years old

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
BMI (Body Mass Index) | 5 Days
  Body Fat, Total Body Water, Muscle Mass, Bone Mass, BMI, calorie, and visceral fat.

SECONDARY OUTCOMES:
Weight | 1 Day
  Body Weight

CONTACTS AND LOCATIONS:
Overall Officials: Guoqing Li, Director, Principal Investigator — Wuhou District Hospital
Locations (1):
- Wuhou District Hospital, Chengdu, Sichuan, China